CLINICAL TRIAL: NCT00115739
Title: Phase II Trial Evaluating Gleevec (Imatinib Mesylate Formerly Known as STI571) in Patients With Anaplastic Thyroid Cancer
Brief Title: Trial Evaluating Gleevec in Patients With Anaplastic Thyroid Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed early due to slow accrual
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Principal Investigator, Francis (Frank) Worden, Principal Investigator, University of Michigan Rogel Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2003-044; IRBMED number 2003-0701 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2005-06-23; First posted 2005-06-24 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Thyroid Cancer
Keywords: Anaplastic Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Carcinoma, Anaplastic | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imatinib (Experimental): Patients will be treated with Imatinib (Gleevec) 400 mg two times a day for eight weeks after which radiologic imaging will be obtained to assess response. Patients who attained a complete response will be treated with four additional weeks of Imatinib. Patients who attain a partial response or stable disease will be treated until a complete response is attained, or until disease progression. All patients with progression of disease will be taken off the study. Patients continuing on the study, will undergo radiologic imaging every eight weeks following their initial response assessment. All patients will be followed until death.
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Imatinib 400 mg capsules were administered twice daily with food for 4 week cycles.
  Other Names: Gleevec

SUMMARY:
Anaplastic thyroid cancers are rare, aggressive tumors. Standard treatment options include surgery and chemoradiation. Few treatment options are available once metastases develop. Recent data suggest that Imatinib (Gleevec) may be advantageous in this patient population. Patients who have been treated for anaplastic thyroid cancer with chemoradiation or surgery who develop recurrent or metastatic disease outside of the field of radiation are eligible. Patients will be treated with Imatinib 400 mg two times a day for eight weeks, followed by radiologic assessment. Patients will be treated until disease progression or a complete response is obtained.

DETAILED DESCRIPTION:
Anaplastic thyroid carcinomas (ATC) are high grade neoplasms, which account for approximately 2% to 5% of primary malignant thyroid tumors but more than 50% of thyroid cancer deaths. Because therapies for anaplastic thyroid carcinoma are very limited with even early stage disease, new approaches for treating this devastating cancer are needed. Recently, imatinib mesylate (Gleevec®), formerly known as STI571, has been approved for the treatment of chronic myelogenous leukemia and for treatment of gastrointestinal stromal tumors, expressing the c-Kit tyrosine kinase. Imatinib is also an inhibitor of the receptor tyrosine kinases for platelet-derived growth factor (PDGF) and stem cell factor, c-Kit, and inhibits PDGF- and SCF-mediated cellular events. Recent data suggest that many if not most, anaplastic thyroid cancers express PDGF receptors, and that these receptors are functional. Additional preclinical work from Japan demonstrates that c-Abl is overexpressed in p53 mutated/deficient anaplastic thyroid carcinoma cell lines and that select inhibition of c-Abl activity by STI571 has a dramatic cytostatic effect in these cells.

Additional data suggest that many, if not most, anaplastic thyroid cancers express PDGF receptors, and that these receptors are functional. Since activation of PDGF receptors is associated with the growth of other tumors and c-Abl is overexpressed in p53-mutated anaplastic thyroid carcinoma cell lines, it seems appropriate to test Gleevec as a therapy for patients with anaplastic thyroid cancer. The specific hypothesis to be tested is that anaplastic thyroid cancers that overexpress PDGF receptors or Abl will respond to Gleevec therapy. The lack of any accepted efficacious therapies for anaplastic thyroid cancer, the poor prognosis of this cancer, and the relatively low toxicity of Gleevec justify this proposed trial.

Patients with anaplastic thyroid carcinoma who are status post best local control with surgery/chemoradiation, who have measurable disease outside their previous field of radiation, are eligible.

The Primary Objective of this study is:

1. To determine the overall response (complete and partial response) rates of patients with anaplastic thyroid cancer treated with Gleevec at the first response assessment (i.e. 8 weeks following the start of Gleevec), following best local control with surgery or radiation/chemoradiation.

The Secondary Objectives include:

1. To measure the grade III/IV toxicities experienced by patients with anaplastic thyroid cancer who are treated with Gleevec.
2. To determine the time to obtain complete or partial responses in patients with anaplastic thyroid cancer treated with Gleevec, following best local control with surgery or radiation/chemoradiation.

Treatment Plan:

Patients will be treated with Imatinib (Gleevec) 400 mg two times a day for eight weeks after which radiologic imaging will be obtained to assess response. Patients who attained a complete response will be treated with four additional weeks of Imatinib. Patients who attain a partial response or stable disease will be treated until a complete response is attained, or until disease progression. All patients with progression of disease will be taken off the study. Patients continuing on the study, will undergo radiologic imaging every eight weeks following their initial response assessment. All patients will be followed until death.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed anaplastic thyroid carcinoma, who have measurable disease.
* Patients with brain metastases are eligible if they have been stable for at least six weeks post-radiation therapy.
* Age 18 years, male or female.
* Karnofsky performance status (KPS) of > 70%.
* Life expectancy of at least 12 weeks.
* Hematologic: ANC 1,500 mm3, hemoglobin 8.0 g/dl, platelets 100,000/mm3
* Normal serum calcium level within normal limits for the institution documented within 14 days prior to registration.
* All patients (including those with liver metastases) must have adequate hepatic function as defined by a serum bilirubin 1.5 x the institutional upper limit of normal (ULN), and ALT and AST <2.5 x ULN, obtained within 14 days prior to registration.
* Patients must have a serum creatinine less than 1.5 x the institutional upper limits of normal (adjusted for age) within 14 days of registration.
* Women of childbearing potential must have a negative pregnancy test at baseline, prior to receiving any study drug. (Pregnant or lactating patients are excluded.)
* Patients of reproductive potential must practice effective contraception while on study and for at least six months after receiving the last dose of study drug.
* All patients must sign an informed consent prior to enrollment.
* No prior history of non-thyroid malignancy, except adequately treated skin cancer or in situ cervical carcinoma or any other cancer in complete remission for at least two years.
* Prior chemotherapy, chemoradiation, radiation therapy, or surgery must have been completed at least 28 days prior to registration, and all toxicities must have resolved. Patients who have been treated with nitrosourea or mitomycin C must be off of these drugs for at least 6 weeks prior to registration.
* Patients must be able to take oral medications.

Exclusion Criteria:

* Anaplastic thyroid cancer that does not overexpress PDGF receptors or c-Abl by immunohistochemistry
* Any medical or psychiatric illness which, in the opinion of the principal investigator, would compromise the patient's ability to tolerate this treatment regimen.
* No concurrent radiotherapy (to the primary tumor) or chemotherapy may be given to the patient during the administration of the study drug.
* Pregnant or lactating women, women of childbearing potential with either a positive pregnancy test (PPT) at baseline, or sexually active females not using reliable contraceptive methods while on study and for at least six months after chemotherapy. (Postmenopausal women must have been amenorrheic for least 12 months to be considered of non-childbearing potential).
* Sexually active males not using reliable contraceptive methods while on the study and for at least six months after chemotherapy.
* Patients with malabsorption syndromes will be excluded.
* Serious concurrent infections.
* Patients who have had previous organ allografts will be excluded.
* Prisoners.
* Patients with chronic liver disease (i.e chronic active hepatitis and cirrhosis).
* Patients with a known diagnosis of human immunodeficiency virus (HIV) infection.
* Patients who have had major surgery within 2 weeks of study entry.
* Patients with grade III/IV cardiac problems as defined by the New York Heart Association Criteria (i.e. congestive heart failure, myocardial infarction within 6 months of study entry).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2004-02; Primary Completion 2008-05 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis P Worden, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants at the Comprehensive Cancer Center outpatient Oncology Clinics at the University of Michigan Health Systems were approached with a brief discussion of the study. If interested, a more detailed discussion of the risks & benefits of the study took place with the subject as well as any family members that may have been present.
Groups:
- Imatinib (Gleevec) Tablets: 4 (100 mg tablets) = 400 mg dose twice per day (morning and evening) for 16 weeks
Period: Overall Study
Arm/Group | Imatinib (Gleevec) Tablets
Started | 11
Completed | 8
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: 11 patients with Anaplastic thyroid cancer were enrolled and were started on imatinib.
Groups:
- Imatinib (Gleevec) Tablets: patients with Anaplastic thyroid cancer were administered Gleevec tablets From February 2004 to May 2007
Arm/Group | Imatinib (Gleevec) Tablets
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (Complete and Partial Response) Rate at 8 Weeks
Description: The number of patients with Complete Response (CR), Partial Response (PR) and Stable Disease (SD) were determined at 8 weeks.
Time Frame: 8 weeks
Population: Eight patients completed 8 weeks of imatinib and were considered evaluable for response.
Measure: Number; unit: participants
Groups:
- Imatinib (Gleevec) Tablets: Subjects were administered oral Gleevec tablets, then tumor response was assessed
Arm/Group | Imatinib (Gleevec) Tablets
Number analyzed (Participants) | 8
participants
  Number of Participants with CR | 0 [9 to 65]
  Number of Participants with PR | 2
  Number of Participants with SD | 4

2. Secondary Outcome: Rate of Grade 3, Grade 4 and Grade 5 Toxicities Experienced by Patients With Anaplastic Thyroid Cancer Who Are Treated With Gleevec
Description: Number of grade 3, grade 4 and grade 5 toxicities experienced by patients with anaplastic thyroid cancer who are treated with Gleevec.
Time Frame: Up to 30 days post treatment
Population: Patients receiving at least one dose of imatinib were included in toxicity analysis.
Measure: Number; unit: events
Arm/Group | Imatinib (Gleevec) Tablets
Number analyzed (Participants) | 11
events
  Number of Grade 3 Toxicities Reported | 29
  Number of Grade 4 Toxicities Reported | 0
  Number of Grade 5 Toxicities Reported | 0

3. Secondary Outcome: 6 Month Progression Free Survival Rate
Description: The percentage of patients with 6 months progression-free survival was estimated. Progression is defined, using RECIST, as a measurable increase in the smallest dimension of any target or non-target lesion, the appearance of new lesions, or the significant clinical deterioration related to progression of patient's disease.
Time Frame: 6 months
Population: Eight patients completed 8 weeks of imatinib and were considered evaluable for response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Imatinib (Gleevec) Tablets
Number analyzed (Participants) | 8
percentage of patients | 27 [7 to 54]

4. Secondary Outcome: 6 Month Survival Rate
Description: The percentage of patients still alive at 6 months was estimated.
Time Frame: 6 months
Population: Eight patients completed 8 weeks of imatinib and were considered evaluable for response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Imatinib (Gleevec) Tablets
Number analyzed (Participants) | 8
percentage of patients | 46 [17 to 71]

ADVERSE EVENTS:
Arm/Group | Imatinib (Gleevec) Tablets
Serious Adverse Events (participants affected / at risk) | 6/11
Other Adverse Events (participants affected / at risk) | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib (Gleevec) Tablets (N=11)
Neuropathy (Nervous system disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Melena / GI Bleeding (Gastrointestinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Ear and labyrinth disorders) | 1 (1)
Syndrome, Other (General disorders) | 2 (3)
Infection Without Neutropenia (Infections and infestations) | 1 (2)
Pericarditis (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib (Gleevec) Tablets (N=11)
Lymphopenia (Investigations) | 6 (19)
Anemia (Blood and lymphatic system disorders) | 6 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Weight Loss (Investigations) | 3 (5)
Fatigue (General disorders) | 7 (18)
Infection (Infections and infestations) | 3 (7)
Skin Rash (Skin and subcutaneous tissue disorders) | 3 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 3 (4)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphasia (Gastrointestinal disorders) | 2 (6)
Nausea (Gastrointestinal disorders) | 5 (7)
Melena / GI Bleeding (Gastrointestinal disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 3 (5)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (10)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary Urgency (Renal and urinary disorders) | 2 (3)
Edema (General disorders) | 7 (14)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Elevated Creatinine (Investigations) | 2 (7)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (8)
Abnormal Aspartate Aminotransferase (AST) (Investigations) | 4 (11)
Hypertension (Cardiac disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
Blurry Vision (Eye disorders) | 2 (2)
Memory Loss (Nervous system disorders) | 2 (2)
Mood Change - Anxiety (Psychiatric disorders) | 1 (1)
Mood Change - Depression (Psychiatric disorders) | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Creatinine Phosphokinase (CPK) (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Depressed Level of Consciousness (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (6)
Fever (General disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (11)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (4)
Incontinence (Renal and urinary disorders) | 1 (1)
Inner Ear / Hearing (Ear and labyrinth disorders) | 1 (3)
Insomnia (Psychiatric disorders) | 1 (1)
Leukopenia (Investigations) | 4 (16)
Lipase (Investigations) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4 (7)
Pain - Other (General disorders) | 5 (5)
Partial Thromboplastin Time (PTT) (Investigations) | 2 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (2)
Rigors / Chills (General disorders) | 2 (2)
Abnormal Alanine Transaminase (ALT) (Investigations) | 4 (5)
Sexual / Reproductive Function (Reproductive system and breast disorders) | 1 (1)
Supraventricular Arrhythmias (Cardiac disorders) | 1 (2)
Sweating (General disorders) | 1 (1)
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Vomiting (Gastrointestinal disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
Study was closed early due to slow accrual. Planned accrual was 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No